CLINICAL TRIAL: NCT04125771
Title: Diclofenac Potassium Alone Versus Diclofenac Potassium With Hyoscine-N-butyl Bromide (HBB in Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aljazeera Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Researcher , lecturer ,Obstetrics and Gynecology , National Research Centre, Aljazeera Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Diclofenac potassium
Record Dates: First submitted 2019-10-11; First posted 2019-10-14 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Hysteroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diclofenac + HBB (Other): Women who will receive Diclofenac + HBB
  Interventions: Diagnostic Test: Diclofenac + HBB with hysteroscopy; Diagnostic Test: Diclofenav + placebo
- Diclofenav + placebo (Other): Women who will receive Diclofenav + placebo
  Interventions: Diagnostic Test: Diclofenac + HBB with hysteroscopy; Diagnostic Test: Diclofenav + placebo

INTERVENTIONS:
Diagnostic Test: Diclofenac + HBB with hysteroscopy — Giving Diclofenac + HBB with hysteroscopy
Diagnostic Test: Diclofenav + placebo — Giving Diclofenac + placebo with hysteroscopy

SUMMARY:
Diclofenac is a proven, commonly prescribed nonsteroidal anti-inflammatory drug (NSAID) that has analgesic, anti-inflammatory, and antipyretic properties, and has been shown to be effective in treating a variety of acute and chronic pain and inflammatory conditions.

DETAILED DESCRIPTION:
Diclofenac is a proven, commonly prescribed nonsteroidal anti-inflammatory drug (NSAID) that has analgesic, anti-inflammatory, and antipyretic properties, and has been shown to be effective in treating a variety of acute and chronic pain and inflammatory conditions.

. As with all NSAIDs, diclofenac exerts its action via inhibition of prostaglandin synthesis by inhibiting cyclooxygenase-1 (COX-1)

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients indicated for diagnostic hysteroscopy including infertility, bleeding, suspected intrauterine pathologies (eg polypi , septea) 2. Reproductive age 20 - 40yrs

Exclusion Criteria:

* 1. Menopausal and amenorrhic patients 2. Contraindication to office hysteroscopy such as:- pelvic inflammatory disease, marked cervical stenosis, pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female who will undergo hysteroscopy
Enrollment: 64 (Actual)
Dates: Start 2020-02-16 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
The number of women who will not feel pain | within half an hour
  the effect of medications on pain sensation

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Study Chair — Algezeera hospitaland National Research Centre ,Egypt
Locations (1):
- Algazeerah and Kasralainy hospital, Giza, Egypt